CLINICAL TRIAL: NCT07133269
Title: Effectiveness of A Care Coach-led Integrated Palliative Surgical Oncology and Rehabilitation Care Model in Patients With Advanced Cancer Undergoing Major Surgery: A Randomized Controlled Trial
Brief Title: Care Coach-led Integrated Palliative Surgical Oncology and Rehabilitation Care Model for Advanced Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Cancer Centre, Singapore (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PHRGOC24jul-0008
Record Dates: First submitted 2025-08-06; First posted 2025-08-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer
Keywords: Palliative Care; Advancer cancer; Cancer rehabilitation; Surgical Oncology; Care coach; Quality of Life
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Patients will receive the current standard of care based on their surgeon's usual clinical practice. [Note: All surgeons in the Division of Surgery & Surgical Oncology (DSSO)- SGH and NCCS are required to attend a basic palliative care course.]
- Care Coach-led Palliative Surgical Oncology (PSO) (Experimental): Patients will receive the current standard of care based on their surgeon's usual clinical practice and the Care Coach-led Palliative Surgical Oncology (PSO) intervention.
  Interventions: Other: Care Coach-led Palliative Surgical Oncology (PSO)
- Care Coach-led Palliative Surgical Oncology with Rehabilitation (PSO+R) (Experimental): Patients will receive the current standard of care based on their surgeon's usual clinical practice, PSO intervention and services from a dedicated rehabilitation service (PSO+R).
  Interventions: Other: Care Coach-led Palliative Surgical Oncology (PSO); Other: Rehabilitation

INTERVENTIONS:
Other: Care Coach-led Palliative Surgical Oncology (PSO) — * Patients will receive the current standard of care based on their surgeon's usual clinical practice.
  * Additionally, patients will receive the Care Coach-led Palliative Surgical Oncology (PSO) intervention during all phases of their surgical journey.
    * After pre-surgery consultations, care coaches will conduct Serious Illness Conversations (SIC) and focus on exploration of patients' hopes and worries, critical functions, social setup, and identification of a healthcare proxy. The SIC will also be conducted at 1, 3, 6, 9 and 12 months post-surgery.
    * The Care coach will also screen for psychological and emotional needs using the Distress Thermometer and Problem List (pre-surgery and at 1, 3, 6, 9 &12 months post-surgery). This will help to identify areas requiring palliative interventions such as symptom management or psychosocial support and for follow-up actions to be taken.
    * ACP will also be offered at each timepoint to those who have yet to do so.
  Arms: Care Coach-led Palliative Surgical Oncology (PSO); Care Coach-led Palliative Surgical Oncology with Rehabilitation (PSO+R)
Other: Rehabilitation — • Patients will receive services from a dedicated rehabilitation service comprising of a Rehabilitation Physician, Physiotherapist, and Dietician.
  * Pre-surgery: Patients will be triaged based on their frailty [Clinical Frailty Scale (CFS)], malnutrition risk [Malnutrition Universal Screening Tool (MUST)], and physical function [5-sit-to-stand (5-STS)] and will receive preventive rehabilitation interventions tailored to their functional needs.
  * During surgical admission: The rehabilitation physician will review the progress of patients and refer them to a dietitian if needed. Patients may be followed-up by a rehabilitation physician one-month post-discharge and referred to a physiotherapist if required.
  * Post-surgery: Patients will be screened by care coaches for health needs using the EQ-5D-5L at months 3, 6, 9 & 12 post-surgery who will make referrals to a rehabilitation physician, nurse and psychologist, as needed.
  Arms: Care Coach-led Palliative Surgical Oncology with Rehabilitation (PSO+R)

SUMMARY:
Advanced cancer is a life-limiting condition that can negatively impact quality of life and function. Patients often suffer from physical, emotional, social, spiritual, and decision-making issues. As such, most would benefit from basic palliative care (PC) which includes establishing goals of care through serious illness conversations (SIC), managing basic pain and other symptoms and addressing psychosocial needs, among others. Patients with advanced cancer are also at higher risk of functional decline due to receiving multiple concurrent treatments. Yet, among patients with advanced cancer undergoing major surgery, there has been little consideration of PC and functional needs.

The palliative surgical care model is a care model in which PC educated surgical oncology teams deliver basic PC, allowing sustainable PC provision to an increasing number of patients living with advanced cancer. In a local pilot palliative surgical care model, it was found that a care coach-led palliative surgical oncology (PSO) care model significantly increased palliative care delivery, ensuring more consistent and comprehensive support for patients. In addition, cancer rehabilitation delivered by rehabilitation professionals addresses functional impairments during the cancer journey, restoring and/or maintaining function and improving quality of life. It also plays a preventive role before surgery, a restorative role during treatment, and a supportive role during cancer progression.

Therefore, to address longitudinal PC and functional needs, an integrated care coach-led palliative surgical oncology rehabilitation (PSO+R) care model involving PC-trained care coaches, surgical oncology teams, rehabilitation professionals, supported by specialist palliative care (SPC) physicians who will provide PC and cancer rehabilitation throughout the patient's advanced cancer journey, is proposed.

DETAILED DESCRIPTION:
Advanced cancer is a life-limiting condition that can negatively impact function, quality of life and exerts an excessive strain on caregivers. In Singapore, up to 60% of cancer patients suffer from advanced (stage 3 or 4) cancer at diagnosis and are recipients of resource-intensive and costly life-prolonging treatments including surgery, chemo-, radiation therapy, among others. In fact, approximately 80% of patients with advanced cancer undergo major surgery at some point of their cancer journey. Given their life-limiting cancer, these patients suffer from physical, emotional, social, spiritual, and decision-making issues that can arise near end-of-life. As such, most would benefit from basic palliative care (PC). This includes establishing goals of care through serious illness conversations (SIC), managing basic pain and other symptoms, and addressing psychosocial needs, among others. As they are often recipients of concurrent intensive multi-modality cancer treatments, patients with advanced cancer are also at higher risk of functional decline, and are ten times more likely to experience morbidity or mortality and have a six-fold increase in risks of 30-day emergency readmissions after major surgery as compared to patients without advanced disease. Yet, among patients with advanced cancer undergoing major surgery, there has been little consideration of PC and functional needs, leading to overall poor quality of life.

Palliative surgical care model is a care model in which PC educated surgical oncology teams deliver basic PC, allowing sustainable PC provision to an increasing number of patients diagnosed and living with advanced cancer. In a local pilot palliative surgical care model, it was found that longitudinal PC (as opposed to during the peri-operative period only) and functional needs during the advanced cancer journey were not well-addressed. Additionally, surgeon-led palliative surgical care was not feasible due to time constraints and competing clinical demands. However, it was found that a care coach-led palliative surgical oncology (PSO) care model significantly increased palliative care delivery, ensuring more consistent and comprehensive support for patients. Cancer rehabilitation delivered by rehabilitation professionals addresses functional impairments during the cancer journey and aims to restore and maintain function and improve quality of life. It plays a preventive role before surgery, restorative during adjuvant treatments, and is supportive during cancer progression.

To address longitudinal PC and functional needs, the investigators propose an integrated care coach-led palliative surgical oncology rehabilitation (PSO+R) care model involving PC-trained care coaches, surgical oncology teams, rehabilitation professionals, supported by specialist palliative care (SPC) physicians who will provide PC and cancer rehabilitation throughout the advanced cancer journey. Care coach-led PSO comprises of care coaches who will screen for PC needs, provide basic PC, and trigger referrals to SPC and surgical team when complex needs arise. The cancer rehabilitation team will screen for functional needs and institute tailored interventions. PSO+R care will be implemented before and up to 1 year after surgery. In contrast, usual care, though surgeons may be trained in PC, they are not supported by care coaches nor cancer rehabilitation or SPC teams. They provide standard peri-operative only care without consideration of the unique needs in advanced cancer. The objective of this proposal is to test the incremental effectiveness of care coach-led PSO+R vs PSO only vs usual care in improving health-related quality of life (HRQoL), functional capacity, and PC delivery and determine the cost-effectiveness of PSO+R over the next most costly intervention, among advanced cancer patients undergoing major surgery. To evaluate its effectiveness, the investigators conduct a 3-arm randomized controlled trial comparing outcomes at 6 months in patients receiving PSO+R vs PSO only vs usual care.

ELIGIBILITY:
Inclusion Criteria:

(i) Patients:

1. Aged 21 and above,
2. Diagnosis of advanced cancer, i.e. stage 3 or 4 solid organ cancer or diagnosed with cancer that requires complex surgery,
3. Planned for elective major surgery (Table of Surgical Procedures (TOSP) table code 4 or more or surgery involves more than one surgical discipline,
4. Able to speak and read English or Chinese

(ii) Caregivers:

1. Age 21 and above,
2. Unpaid family or informal caregiver who takes direct care of the patient's day-to-day and healthcare needs, or ensures provision of care to meet the needs, or who is the decision maker with regard to the patient's needs and healthcare,
3. Able to speak and read English or Chinese.

(iii) Healthcare Providers (Qualitative interview only):

1. Age 21 and above,
2. Currently working as a Healthcare professional at SGH or NCCS and involved in this study.

Exclusion Criteria:

(i) Patients:

1. Patient refusal,
2. Have complex PC needs requiring specialty palliative care (SPC) intervention before surgery,
3. Active mental illness or severe dementia and certified unfit to make medical decision by a specialist physician,
4. Scheduled for Emergency surgery.

(ii) Caregivers:

1. Unwilling to participate in the study.

(iii) Healthcare Providers (Qualitative interview only):

1. Unwilling to participate in the Qualitative interview.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-08-20 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
HRQoL in patients post-surgery (measured by FACT-G) | Baseline, 6 months post-surgery
  -The Functional Assessment of Cancer Therapy - General (FACT-G) is a well-validated HRQoL questionnaire that covers 4 domains - physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items) and functional well-being (7 items). Each item has response choices in a 5-point Likert-type scale, with a maximum value of 4 (being, "Very much") and a minimum value of 0 (being "Not at all"). Higher scores indicate a better quality of life.

SECONDARY OUTCOMES:
HRQoL in patients post-surgery (measured by FACT-G) | Baseline, 1, 3, 9 and 12 months post-surgery
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a well-validated HRQoL questionnaire that covers 4 domains - physical well-being (7 items), social/family well-being (7 items), emotional well-being (6 items) and functional well-being (7 items). Each item has response choices in a 5-point Likert-type scale, with a maximum value of 4 (being, "Very much") and a minimum value of 0 (being "Not at all"). Higher scores indicate a better quality of life
HRQoL in patients post-surgery (measured by EQ-5D-5L) | Baseline, 1, 3, 6, 9, 12 months post-surgery
  The 5-level EuroQol-5 Dimension instrument (EQ-5D-5L) is a HRQoL questionnaire with five domains (mobility, selfcare, usual activities, pain/discomfort, anxiety/depression) and has five levels for each domain. Scores from all five items will be used to derive a single utility score ranging from 0 to 1, with 0 representing the worst possible health to 1 representing perfect health. It also contains a health state component and a visual analog scale.
Frailty in patients post-surgery | Baseline, 1, 3, 6, 9 & 12 months post- surgery
  The Clinical Frailty Scale (CFS) is a well-validated scale to screen for frailty. It is a 9-point scale that quantifies the frailty of the individual based on his/her functioning. There is a minimum score of 1 (indicating "Very Fit) and 9 (indicating Terminally Ill). A higher score is indicative of greater frailty.
Functional lower extremity strength, transitional movements, balance, and fall risk in patients post-surgery | Baseline, 1, 3, 6, 9 & 12 months post- surgery
  The Five Times Sit-to-Stand (5-STS) test is a test to assess functional lower extremity strength, transitional movements, balance, and fall risk in patients. The patient is asked to sit against the back of a chair. The time taken to change from a seated position to a standing position five times is measured. A time of less than 12 seconds is linked to better functional lower extremity strength, transitional movements, balance, and reduced risk for falls.
Malnutrition and risk for malnutrition in patients post-surgery | Baseline, 1, 3, 6, 9 & 12 months post- surgery
  The Malnutrition Universal Screening Tool (MUST) is a tool to assess for malnutrition and the risk for malnutrition. It consists of five steps and assesses one's risk for malnutrition by evaluating one's Body Mass Index (BMI), rate of weight loss and presence of acute disease. A score of 0 indicates low risk of malnutrition, whereas a score of 2 or more indicates a high risk of malnutrition.
Patient-surgeon relationship post-surgery | Baseline, 1-month post-surgery
  The Human Connection (THC) scale measures the therapeutic alliance between patients and their physicians. It consists of 16 questions. Each item has response choices in a 4-point Likert-type scale, with a maximum value of 4 and a minimum value of 1. Higher scores indicate a stronger patient-surgeon relationship.
Documentation of Serious Illness Conversations (SIC) with patients pre-surgery | Baseline (i.e pre-surgery)
  Serious Illness Conversations (SIC) (adapted from Ariadne Labs) enable Healthcare providers to understand patients' values and goals. This would be used as part of a palliative care delivery quality indicator.
Establishment of Advance Care Planning with patients | Within 1-year post-surgery
  Advance Care Planning is a process of discussing one's values and future care preferences. This would be used as part of a palliative care delivery quality indicator.
Patients' receipt of specialist palliative care, when complex palliative care needs arise. | Within 1-year post- surgery
  Patients with complex palliative care needs will be referred to specialist palliative care physicians, meeting the needs of patients and promoting HRQoL. This would be used as part of a palliative care delivery quality indicator.
Healthcare utilization of patients | Up to 1-year post-surgery
  Healthcare utilization will be determined by extracting the length of index hospitalization, all-cause emergency department visits, and total hospital days up to 1-year post-surgery.
Cost of intervention(s) | Up to 1-year post-surgery
  Inpatient and outpatient billing records will be considered in total all-cause healthcare costs up to 1-year post-surgery.
Cost-effectiveness of intervention(s) | Up to 1-year post-surgery
  The incremental cost-effectiveness of PSO and PSO+R will be quantified from the health system perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Jolene Wong, MBBS, MMed (Surgery), MPH, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - National Cancer Centre Singapore, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No